CLINICAL TRIAL: NCT01320124
Title: Knee Joint Contractures: Reversibility and Molecular Pathways
Brief Title: Creating a Tissue Bank of Knee Capsules
Status: Withdrawn | Type: Observational
Sponsor: Ottawa Hospital Research Institute (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government)
Responsible Party: Principal Investigator, Dr. Guy Trudel, Researcher, Ottawa Hospital Research Institute
Other Study IDs: 2010930-01H
Record Dates: First submitted 2011-03-18; First posted 2011-03-22 (Estimated); Last update posted 2015-04-23 (Estimated); Status verified 2015-04

CONDITIONS: Osteoarthritis; Knee Joint Contractures
Keywords: Contractures; Total knee arthroplasty; Tissue bank; Osteoarthritis; Gene expressions
MeSH Terms: conditions — Osteoarthritis; Contracture

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — A blood sample will be drawn from each subject and stored with the capsule tissue.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- osteoarthritis, total knee arthroplasty: The main cohort will have a total knee arthroplasty and will not develop a contracture post surgery. We will analyze differntial gene expression in all subjects.
- contracture post arthroplasty: A small group (1.3%) will develop a contracture post total knee arthroplasty. A second sample will be taken at the time of corrective surgery. The 2 samples will be compared for gene expression in the same subject. This group will also be compared to the main cohort for differential gene expression.

SUMMARY:
A contracture is a pathological condition limiting range and function of joints. Contractures of large and small joints alike will affect one's ability to independently perform daily activities such as eating, dressing or walking. Current treatments for contractures include physical stretching, the use of assistive devices or, rarely, surgery. Despite prolonged treatments, patients with contractures rarely regain complete mobility. Progress in preventing and treating contractures will be possible only through an understanding of the biological and molecular processes involved. Our group has established and validated an animal model to study the histological events and the molecular mechanisms involved in joint contractures. We have provided evidence for capsule stiffness, characterized cartilage degeneration, and identified four genes whose expression is altered in the cartilage of a knee joint with contracture. The work we propose in the current study aims at finding genes and pathways in the joint capsule associated with knee joint contractures. The results will identify new avenues for treating the large number of patients suffering from contractures.

DETAILED DESCRIPTION:
We propose to constitute a bank of capsule samples from people with osteoarthritis undergoing primary total knee arthroplasty. It is expected that about 1.3% of people will develop a contracture post arthroplasty. A second sample will be taken from those that require surgery for release of contracture or revision. We will study histological characteristics and compare gene expression between the primary sample and the contracture sample in the same patient. In order to determine whether intrinsic genetic factors influence the develpment of joint contractures in the osteoarthritis population, all specimens will be analyzed for differential gene expression between patients with and without knee contractures post arthroplasty.

The remaining capsule tissue not used for this study will be banked and made available to other researchers.

ELIGIBILITY:
Inclusion Criteria:

* Osteoarthritis, booked for a total knee arthroplasty

Exclusion Criteria:

* Transmissible disease (e.g., HIV infection, hepatitis B or C)
* Suspected neoplasia
* Suspected infection (which can cause arthrofibrosis)
* Hypertrophic scarring

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients booked for a total knee arthroplasty at the Ottawa Hospital, with a primary diagnosis of osteoarthritis.
Sampling Method: Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2011-03; Primary Completion 2015-04 (Actual); Study Completion 2015-04 (Actual)

PRIMARY OUTCOMES:
development of contracture post total knee arthroplasty | Within 1 year
  1.3% of subjects are expected to develop a contracture post toal knee arthroplasty within a year of the surgery.

CONTACTS AND LOCATIONS:
Overall Officials: Guy Trudel, MD, Principal Investigator — University of Ottawa
Locations (1):
- The Ottawa Hospital, Ottawa, Ontario, Canada